CLINICAL TRIAL: NCT04578379
Title: Interest of the IRAP (Insulin Regulated Amino Peptidase) Marker to Assess the Levels of Insulin Resistance in a Cohort of Insulin-resistant Subjects Due to DUNNIGAN Lipodystrophy
Brief Title: Insulin Regulated Amino Peptidase in Patients With Familial Lipodystrophy of DUNNIGAN
Acronym: IRAP-DUN
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de la Réunion (Other)
Responsible Party: Sponsor
Other Study IDs: 2017/CHU/07
Record Dates: First submitted 2020-10-01; First posted 2020-10-08 (Actual); Last update posted 2020-10-08 (Actual); Status verified 2020-10

CONDITIONS: Lipodystrophy; Insulin Resistance
MeSH Terms: conditions — Lipodystrophy; Insulin Resistance

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Familial Partial Lipodystrophy type 2 (FPLD2) is a heterogeneous group of rare lipodystrophy due to autosomal dominant mutation in LMNA encoding Lamin A/C. Lamins A and C form with the B-type lamins the lamina network underlying the nuclear envelope. Lamins are major components that provide structural and mechanical stability for the nucleus ubiquitously. Lamins are also key epigenetic regulator. Mutations in LMNA are involved in different inherited pathologies as Emery-Dreifuss muscular Dystrophy, Limb Girdle muscular dystrophy, dilated cardiomyopathy and conduction system disease, Charcot Marie Tooth Disorder type 2, mandibuloacral dysplasia, Hutchinson Gilford progeria and Dunnigan-type-familial partial lipodystrophy (FPLD2).

Inherited lipodystrophy prevalence is reported around 1.3 to 10 cases per million worldwide and FPLD2 is the most frequent of all. Nevertheless, recent reports with systematic screening in all non-obese patients with type 2 diabetes or metabolic syndrome found higher prevalence of lipodystrophy up to 1/7000 subjects. FPLD2 remain a rare group of disease and only relatively small and heterogeneous cohorts of patients are reported. For this reason it is difficult to fully decipher all aspects of this rare group of diseases. The "typical" FPLD2 is associated with missense mutation affecting the arginin residue in position 482 (p.R482Q,p.R482W,p.R482L). Patients harbouring mutation in other spot are considered to have "atypical" lipodystrophy. The "typical" FPLD2 start around puberty with progressive subcutaneous fat loss in upper limbs, gluteo-femoral adipose tissue and trunk and fat accumulation in the cervicofacial area, neck, upper trunk, labia majora and visceral fat. Resulting from the inability to store fat, patients affected by inherited lipodystrophy develop severe metabolic syndrome and its complications: type 2 diabetes (DT2), dyslipidaemia, nonalcoholic fatty liver disease (NAFLD) and premature cardiovascular disease (CVD).

In 2006 a specific mutation of LMNA has been described in a patient originated from La Réunion living in France mainland. To date this mutation have only been reported in patient native from La Réunion and is called 'Reunionese' mutation and consist in a G insertion after nucleotide 5670 (codon 654) in the prelamin-A-specific exon 11 (g.5670_5671insG) p.T655fsX49 that lead to a longer and non farnelysated prelamin A lacking the C-terminal CSIM motif. As a result, nonfarnelysated mutated prelamin A accumulated in the cells leading to oxidative stress and premature cell senescence. The 'Reunionese' mutation is expressed in 2 forms either homozygous or heterozygous. Homozygous patients present with more severe phenotype and cardiac laminopathy.

The aim of our study is to update the characterization of the patients diagnosed with the 'Reunionese' mutation. The investigators report here the largest cohort of patient with FPLD2 due to one single LMNA mutation either homozygous or heterozygous.

DETAILED DESCRIPTION:
The investigators systematically reviewed the medical records of patients with a diagnosis of genetically confirmed FPLD at Reunion University Hospital (La Réunion, France) from 2006 (beginning of the screening for lipodystrophy) to 2020. Due to the high prevalence of lipodystrophy in our island and to follow the recommendations in follow up, a specific check-up is organized in our centre since 2016. For this study the investigators collected the data from patients who carried the same LMNA 'Reunionese' mutation: p.T655fsX49 and who benefited a complete check-up in our centre since 2016. Between 2006 and 2020, 97 patients were diagnosed with FPLD at Reunion University Hospital. Three different mutations were diagnosed: 85 subjects carried the 'Reunionese' mutation LMNA p.T655fsX49 (70 heterozygous and 15 homozygous), 8 carried the mutation LMNA p.R582H and 3 subjects carried a mutation of PPARγ. Among the carrier of the mutation LMNA p.T655fsX49, 70 subjects benefit a recent follow up with complete examination (61 heterozygous (HTZ) and 9 homozygous (HMZ)) and 4 deceased (all carrier of the homozygous form).

ELIGIBILITY:
Inclusion Criteria:

* Adult subject with homozygous or heterozygous partial Dunnigan lipodystrophy
* Informed consent siged by the subject

Exclusion Criteria:

* Hemoglobin level <7 mg / dl or <9-10 mg / dl for patients with cardiovascular or respiratory pathology.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with partial lipodystrophy from DUNNIGAN and benefiting from regular monitoring and an annual assessment of the impact of their pathology at the Reunion University Hospital
Sampling Method: Non-Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2020-03-01 (Actual); Study Completion 2020-07-01 (Actual)

PRIMARY OUTCOMES:
IRAP assay | between day 7 and day 15
  To assess the value of the IRAP assay for assessing the level of insulin resistance in a cohort of patients with Dunnigan syndrome of different severity.

CONTACTS AND LOCATIONS:
Overall Officials: Estelle NOBECOURT, MD, Principal Investigator — Centre Hpospitalier Universitaire de La REUNION
Locations (1):
- Centre Hospitalier Universitaire de La Réunion, Saint-Pierre, Reunion

IPD SHARING:
Plan to Share IPD: No